CLINICAL TRIAL: NCT03100188
Title: Designer Dialysis: Designing a Peritoneal Dialysis Prescription That Fits a Patient's Lifestyle
Brief Title: Designer Dialysis Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Mihran Naljayan, principal investigator, Louisiana State University Health Sciences Center in New Orleans
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#9421
Record Dates: First submitted 2017-03-12; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Peritoneal Dialysis; Quality of Life
Keywords: peritoneal dialysis; incremental peritoneal dialysis; quality of life; end stage renal disease; adequacy
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: one cohort of patients who meet inclusion criteria had intervention and followed for 12 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- modified PD (Experimental): Patients with residual renal kt/v were placed in intervention group
  Interventions: Other: modified PD prescription

INTERVENTIONS:
Other: modified PD prescription — For patients on CAPD, fewer daily exchanges or fewer total weekly exchanges are prescribed. Patients on CCPD are prescribed shorter cycler time or fewer total cycles during the week.

SUMMARY:
This study aims to use modified peritoneal dialysis prescriptions to achieve adequate clearance and volume removal while decreasing the number of exchanges or time spent on dialysis, evaluating maintenance of residual renal function, and improving quality of life.

DETAILED DESCRIPTION:
Patient's currently on peritoneal dialysis at our program can be considered for this study. In order to be enrolled, patients patient's must have significant residual renal function defined as a renal Kt/V >1.0. These patients will then be consented, and if agreeable, the participant's dialysis prescriptions will be modified to decrease their peritoneal dialysis. For patients on continuous ambulatory peritoneal dialysis (CAPD), this may mean less exchanges in a 24 hour period, or less exchanges over the course of the week (does not need to perform exchanges every day). Patients who are continuous cycler peritoneal dialysis (CCPD) will be modified to shorter cycler times, or also less cycles during the course of the week (does not need cycler therapy every day).

Patients will need to continue achieving adequate weekly total Kt/V of greater than or equal to 1.7 as per national recommendations and the clinical guidelines within our unit. This is calculated using the residual renal (RR) Kt/v and the PD Kt/V. Patients will also perform monthly 24 hour urine collections for urinary volume, creatinine clearance, and urea clearance. Adequacy is typically measured every 3 months based on our internal lab requirements, but patients will need to perform adequacy measurements any time their prescription is changed. The investigators will measure monthly labs per routine including albumin, parathyroid hormone (PTH), serum phosphorus, and hemoglobin.

The investigators hypothesize that patients will have a better quality of life (QoL) while on a modified dialysis prescription with less exchanges or less cycler time as assessed by the kidney disease quality of life (KDQOL-36) survey tool. The investigators believe that patients with higher levels of residual renal function (≥ 2 mL/min) can perform fewer peritoneal dialysis exchanges while still achieving and maintaining adequate clearance of solute and appropriate volume removal. The investigators also believe that by maximizing the use of the residual renal function, the investigators can adjust the peritoneal dialysis prescription by decreasing the numbers of manual exchanges per day, decreasing cycler time, or possibly decreasing the number of days of dialysis each week. With the benefit of less dialysis time or exchanges per day, the investigators believe patients will have a decreased "burnout" rate by allowing them to have a better QoL and not feel burdened by the dialysis therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients on either CAPD or CCPD and had both residual renal (RR) Kt/V ≥ 1.0 and total Kt/V values ≥ 1.7.

Exclusion Criteria:

* patients who did not meet the values of RR Kt/V and total Kt/V specified above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
change in quality of life | at the time of enrollment and again after 12 months
  change in survey results of modified KDQOL 36 survey

SECONDARY OUTCOMES:
change in residual renal kt/v | 30 days after enrollment, and then every 3 months for a total of 12 months after enrollment.
  change in RR kt/v
change in PD Kt/V | 30 days after enrollment, and then every 3 months for a total of 12 months after enrollment.
  change in PD Kt/V
change in total kt/v | 30 days after enrollment, and then every 3 months for a total of 12 months after enrollment.
  change in total kt/v; this is calculated by adding RR kt/v and PD kt/v
change in serum albumin | monthly for 12 months after enrollment
  change in serum albumin level
change in 24 hour urine output | monthly for 12 months after enrollment
  change in 24 hour urine output

CONTACTS AND LOCATIONS:
Overall Officials: Mihran Naljayan, MD, Principal Investigator — LSU School of Medicine

IPD SHARING:
Plan to Share IPD: No